CLINICAL TRIAL: NCT01473680
Title: Pilot Study of Neuropsychologic and Electrophysiological Features of Cancer-Related Cognitive Side Effects in Racial and Ethnic Minority Breast Cancer Patients
Brief Title: Neuropsychologic and Electrophysiological Features of Cancer-Related Cognitive Side Effects in Racial and Ethnic Minority Breast Cancer Patients
Status: Terminated | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The City College of New York (Other); Ralph Lauren Center for Cancer Care and Prevention (Other); Lincoln Medical and Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-139
Record Dates: First submitted 2011-11-10; First posted 2011-11-17 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: minority breast cancer patients; EEG; Evaluation; Questionnaires; 11-139
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Patients who will receive chemo: This study is an assessment of individuals' cognitive functioning through administration of NP and psychological instruments and EEG. These assessments do not require manipulation of a participant's environment to elicit change in behavior or treatment outcome. NP and psychological instruments.
  Interventions: Other: EEG, Neuropsychological Evaluation, Psychological Questionnaires, Medical Questionnaire
- Patients who will not receive chemo: This study is an assessment of individuals' cognitive functioning through administration of NP and psychological instruments and EEG. These assessments do not require manipulation of a participant's environment to elicit change in behavior or treatment outcome. NP and psychological instruments.
  Interventions: Other: EEG, Neuropsychological Evaluation, Psychological Questionnaires, Medical Questionnaire
- Healthy Controls: This study is an assessment of individuals' cognitive functioning through administration of NP and psychological instruments and EEG. These assessments do not require manipulation of a participant's environment to elicit change in behavior or treatment outcome. NP and psychological instruments.
  Interventions: Other: EEG, Neuropsychological Evaluation, Psychological Questionnaires, Medical Questionnaire

INTERVENTIONS:
Other: EEG, Neuropsychological Evaluation, Psychological Questionnaires, Medical Questionnaire — Participants will complete a medical/psychiatric history questionnaire, and a standardized battery of neuropsychological (NP) tests and psychological instruments. EEG recording will be made as participants engage in tasks of basic perceptual or pre-attentive processes and selective attention. Following chemotherapy (and a matched interval for the no-chemotherapy and healthy control groups), the standardized battery of NP tests, psychological instruments, and EEG will be repeated.
  Groups: Patients who will receive chemo
Other: EEG, Neuropsychological Evaluation, Psychological Questionnaires, Medical Questionnaire — Participants will complete a medical/psychiatric history questionnaire, and a standardized battery of neuropsychological (NP) tests and psychological instruments. EEG recording will be made as participants engage in tasks of basic perceptual or pre-attentive processes and selective attention. Following chemotherapy (and a matched interval for the no-chemotherapy and healthy control groups), the standardized battery of NP tests, psychological instruments, and EEG will be repeated.
  Groups: Patients who will not receive chemo
Other: EEG, Neuropsychological Evaluation, Psychological Questionnaires, Medical Questionnaire — Participants will complete a medical/psychiatric history questionnaire, and a standardized battery of neuropsychological (NP) tests and psychological instruments. EEG recording will be made as participants engage in tasks of basic perceptual or pre-attentive processes and selective attention. Following chemotherapy (and a matched interval for the no-chemotherapy and healthy control groups), the standardized battery of NP tests, psychological instruments, and EEG will be repeated.
  Groups: Healthy Controls

SUMMARY:
This study is being done to find out if it is possible to enroll minority women with breast cancer in a study of how chemotherapy may affect their ability to answer certain questions and perform certain tasks that measure brain activity. The investigators want to look at thinking and brain activity in patients to see if cancer treatments can cause any brain changes. For this study, women without cancer, are being asked to participate in order to compare the answers to the questions and the brain wave activity measured in the women with cancer to women who don't have cancer.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years old, but not older than 61 years old;
* Is female;
* Is Hispanic of any race or Black/African American
* Is fluent in English (see explanation in Section 7.0 Assessment / Evaluation Plan - Language Determination);
* Has a diagnosis of breast cancer (Stage I-III);
* Is treatment naïve and scheduled to receive chemotherapy, radiation, or endocrine therapy.

Healthy Control Subject Inclusion Criteria

* Is at least 18 years old, but not older than 61 years old;
* Is female;
* Is Hispanic or Black Non-Hispanic;
* Is fluent in English

Exclusion Criteria:

* Participants with neurologic illnesses affecting cognition, (i.e., Traumatic Brain Injury with a loss of consciousness >30 min., etc.) or severe psychiatric illness (i.e., schizophrenia, bipolar disorder, etc.);
* A hearing or visual deficit that impairs the ability to participate in the EEG tasks.
* Any condition which prevents application of the 160 EEG electrodes spaced evenly across the participant's scalp, which includes dreadlocks, and hair extensions applied by weaving, braiding, gluing, or clips-. unless the participants are willing to undo these styles prior to the EEG.
* Mini-Mental State Exam (MMSE) <16 (telephone version); MMSE <20 (in-person version)
* Prior chemotherapy for any malignancy
* Regularly taking opiates or take a daily, morning benzodiazepine or have taken a prn benzodiazepine prior to the assessment.

Healthy Control Subject Exclusion Criteria

* Current or historical cancer diagnosis (a previous diagnosis of basal cell skin carcinoma is allowable)
* History of neurologic illnesses affecting cognition, (i.e., Traumatic Brain Injury with a loss of consciousness >30 min., etc.) or severe psychiatric illness (i.e., schizophrenia, bipolar disorder, etc.);
* A hearing or visual deficit that impairs the ability to participate in the EEG tasks.
* Any condition which prevents application of the 160 EEG electrodes spaced evenly across the participant's scalp, which includes dreadlocks, and hair extensions applied by weaving, braiding, gluing, or clips-. unless the participants are willing to undo these styles prior to the EEG
* Mini-Mental State Exam (MMSE) <16 (telephone version); MMSE <20 (in-person version)
* Regularly taking opiates or takes a daily, morning benzodiazepine or has taken a prn benzodiazepine prior to the assessment.

Ages: 18 Years to 61 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: MSKCC clinic, The Ralph Lauren Center for Cancer Care and Prevention (RLCCCP)located in Harlem and Lincoln Hospital located in the Bronx.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
neuropsychologic (NP) features | 2 years
  through administration of NP and psychological instruments and EEG

SECONDARY OUTCOMES:
electrophysiologic features | 2 years
  through administration of NP and psychological instruments and EEG

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ryan, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - The City College of New York, New York, New York
  - Lincoln Hospital, The Bronx, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm